CLINICAL TRIAL: NCT05783349
Title: To Study the Predictive Value of Th1, Th2 and Th17 Cytokine Serum Levels Produced After Non-specific Stimulation on the Success of Embryo Implantation
Brief Title: Predictive Value of Th1, Th2 and Th17 Cytokines on the Success of Embryo Implantation (ImmuNoFertilité)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-PP-17
Record Dates: First submitted 2023-02-10; First posted 2023-03-24 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Assisted Reproduction
Keywords: Repeated Implantation Failure (RIF); Embryo implantation; T cells activation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women treated in the Medically Assisted Procreation (MAP) center of Nice (Other)
  Interventions: Biological: Unique blod sample

INTERVENTIONS:
Biological: Unique blod sample — sampling of 4mL of blood on lithium heparin tube, the day of frozen embryo implantation

SUMMARY:
Infertility affects approximately 10-15% of the population. The number of assisted reproduction procedures has increased by a factor of 3 to 5.3 worldwide over the last 20 years. Despite recent techniques, pregnancy rates seem to be limited to 35% by embryo transfer. Embryo implantation depends on two factors: the quality of the embryo and the endometrial receptivity. Although good quality embryos are transferred, implantation may not occur. Changes in the maternal cytokine profile at the time of implantation may result in poor implantation or early abortions. Consequently, a misdirection of the immunological profile could be responsible for repeated implantation failure (RIF). The definition of RIF is not consensual, but most commonly refers to 3 failures after good quality embryo transfer, and would affect between 5 and 10% of patients.

The possibility of defining a predictive immune profile for RIF from a peripheral blood sample is debated. However, after stimulation of immune cells in peripheral blood, patients with RIF show an excessive pro-inflammatory profile.

Our objective is to assess the activation of T cells and innate immune cells (via an anti-CD3 agonist and a TLR7-8 ligand, respectively) from a blood sample to predict implantation success after frozen embryo transfer. This functional test is easy to use and applicable in a clinical routine.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (aged 18 and above) treated in the Medically Assisted Procreation (MAP) center of the University Hospital of Nice, in the process of a frozen embryo transfer
* Social security affiliation
* Signed consent

Exclusion Criteria:

* Contra-indication to frozen embryo transfer
* Ongoing infection
* Patients under guardianship

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 255 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
Ex vivo comparison of the immune profile between patients with Repeated Implantation Failure and patients with successful implantation. | 24 months
  The immune profiles are defined as the concentrations (in IU/mL or pg/mL) and ratios of proinflammatory and anti-inflammatory cytokines measured after nonspecific stimulation of peripheral blood cells from each patient: IFNγ, IL6, IL1β, TNFα, IL4, IL10, TGFβ, IFNγ/IL4, IFNγ/IL10, IFNγ/TGFβ, IL6/IL4, IL6/IL10, IL6/TGFβ, IL1β/IL4, IL1β/IL10, IL1β/TGFβ, TNFα/IL4, TNFα/IL10, TNFα/TGFβ.

SECONDARY OUTCOMES:
Ex vivo comparison of the immune profile between patients with one implantation failure and patients with successful implantation. | 24 months
  The immune profiles are defined as the concentrations (in IU/mL or pg/mL) and ratios of proinflammatory and anti-inflammatory cytokines measured after nonspecific stimulation of peripheral blood cells from each patient: IFNγ, IL6, IL1β, TNFα, IL4, IL10, TGFβ, IFNγ/IL4, IFNγ/IL10, IFNγ/TGFβ, IL6/IL4, IL6/IL10, IL6/TGFβ, IL1β/IL4, IL1β/IL10, IL1β/TGFβ, TNFα/IL4, TNFα/IL10, TNFα/TGFβ.
Ex vivo comparison of the immune profile between patients with one implantation failure in the context of inflammatory disorder (such as endometriosis) and patients with successful implantation. | 24 months
  The immune profiles are defined as the concentrations (in IU/mL or pg/mL) and ratios of proinflammatory and anti-inflammatory cytokines measured after nonspecific stimulation of peripheral blood cells from each patient: IFNγ, IL6, IL1β, TNFα, IL4, IL10, TGFβ, IFNγ/IL4, IFNγ/IL10, IFNγ/TGFβ, IL6/IL4, IL6/IL10, IL6/TGFβ, IL1β/IL4, IL1β/IL10, IL1β/TGFβ, TNFα/IL4, TNFα/IL10, TNFα/TGFβ.
Ex vivo comparison of the immune profile between patients with a pregnancy failure and patients with an active pregnancy at the end of the first trimester. | 24 months
  The immune profiles are defined as the concentrations (in IU/mL or pg/mL) and ratios of proinflammatory and anti-inflammatory cytokines measured after nonspecific stimulation of peripheral blood cells from each patient: IFNγ, IL6, IL1β, TNFα, IL4, IL10, TGFβ, IFNγ/IL4, IFNγ/IL10, IFNγ/TGFβ, IL6/IL4, IL6/IL10, IL6/TGFβ, IL1β/IL4, IL1β/IL10, IL1β/TGFβ, TNFα/IL4, TNFα/IL10, TNFα/TGFβ.
  Pregnancy test: βhCG concentration on blood sample in IU/L. Result of the ultrasound performed routinely during the first trimester (between 4 and 11 amenorrhea weeks): presence or absence of intrauterine pregnancy , progressive or not.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No
Sharing data is not planned